CLINICAL TRIAL: NCT01860183
Title: Comparison of 3g Versus 2g Mycophenolate Mofetil in Combination With Tacrolimus on Progression of Chronic Histology Changes in Kidney Transplant Recipients
Brief Title: Effect of 3g Versus 2 g MMF in Combination With Tacrolimus on Progression of Renal Allograft Interstitial Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Hospital Merkur (Other)
Collaborators: University Medical Centre Ljubljana (Other); University Hospital Rijeka (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHMerkur
Record Dates: First submitted 2013-05-18; First posted 2013-05-22 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2014-01

CONDITIONS: Kidney Transplantation; Kidney Failure
Keywords: kidney transplantation; chronic allograft dysfunction; mycophenolate mofetil; Chronic
MeSH Terms: conditions — Renal Insufficiency; Bronchiolitis Obliterans Syndrome | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MMF 3g daily (Experimental)
  Interventions: Drug: Mycophenolate mofetil
- MMF 2 g daily (Active Comparator)
  Interventions: Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Mycophenolate mofetil — Mycophenolate will be administered to all study patients at dose of 3 g daily for the first seven days posttransplant. Afterwards, study patients will continue, as randomized, on either 3 g, or 2 g MMF daily.

SUMMARY:
Development of chronic changes (scarring) in transplanted kidney tissue is a major cause of long-term kidney function deterioration and ultimately graft loss. It results from both immunologic and non-immunologic mechanisms. Mycophenolate mofetil (MMF) is immunosuppressive drug used for prevention of rejection after kidney transplant, usually in combination with a calcineurin inhibitor (tacrolimus or cyclosporine), with or without corticosteroids. Besides immunosuppression, MMF may also have direct antifibrotic properties. Tacrolimus has potent immunosuppressive effects and is the cornerstone of contemporary posttransplant immunosuppressive therapy in kidney recipients. However, it is also nephrotoxic. The hypothesis of the present study is that in the setting of similar net immunosuppression, higher dose of MMF (3 g daily) will result in slower progression of kidney fibrosis during first year posttransplant as compared to MMF 2 g daily. To test this hypothesis, the present study will randomly assign low immunological risk kidney transplant recipients to either 2g or 3 g MMF daily, in combination with tacrolimus, with, or without maintenance steroids. All patients will have kidney biopsy at implantation and at 12 months after transplantation. Main outcome will be 1-year change in chronic kidney histology (interstitial fibrosis) assessed by protocol biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. first kidney or kidney-pancreas transplantation
2. CDC PRA <=20%

Exclusion Criteria:

1. dual kidney transplantation
2. AB0 incompatible transplantation
3. 0 biopsy ci, ct, cv, or ah score >=2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Progression of interstitial fibrosis (ci) | 1 year

SECONDARY OUTCOMES:
Estimated glomerular filtration rate | 1 year
Time to first acute rejection episode | up to 1 year
Progression of other chronic scores | 1 year
Graft loss | 1 year
Patient survival | 1 year

OTHER OUTCOMES:
Frequency of infections requiring hospitalization | 1 year
Frequency of CMV viremia | 1 year
Frequency of BK viremia | 1 year
Frequency of BK nephropathy | 1 year
Development of donor-specific antibodies | 1 year
Renal morphology and hemodynamics assessed by ultrasound | 1 year
  Subset of study patients

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Merkur, Zagreb, HR, Croatia

REFERENCES:
- [Derived] Wajih Z, Karpe KM, Walters GD. Interventions for BK virus infection in kidney transplant recipients. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD013344. doi: 10.1002/14651858.CD013344.pub2. PMID 39382091